CLINICAL TRIAL: NCT06334276
Title: Developing an Utstein-style Danish Drowning Registry: Nationwide Fatal and Nonfatal Drowning Data Since 2016
Acronym: DROWN_INHOS
Status: Recruiting | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Principel Investigator, Region Zealand
Other Study IDs: DROWN_INHOS
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Drowning; Drowning, Near; Drowning; Asphyxia; Drowning and Nonfatal Submersion; Drowning or Immersion of Unknown Intent; Drowning and Submersion, Undetermined Intent; Drowning and Submersion While in Bath-Tub; Drowning and Submersion While in Natural Water; Drowning and Submersion While in Swimming-Pool
Keywords: Danish Drowning Formula; Drowning; Danish Prehospital Drowning Data; Registry; Database; Emergency Medical Service; Utstein; Register; Epidemiology
MeSH Terms: conditions — Drowning; Near Drowning; Asphyxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fatal drowning: This group of patients have died before 30 days after the drowning incident.
  Interventions: Other: Drowning
- Non-fatal drowning: This group of patients have survived until 30 days after the drowning incident.
  Interventions: Other: Drowning

INTERVENTIONS:
Other: Drowning — Drowning is defined by the WHO in 2002 as "the process of experiencing respiratory impairment from submersion or immersion in liquid"

SUMMARY:
This nationwide, registry-based study aims to link Danish Prehospital Drowning Data data with inhospital data to develop a Utstein-style Danish Drowning Registry. This study will report mortality and neurological outcomes 30 days after a drowning incident since 2016.

DETAILED DESCRIPTION:
Purpose

The purpose of this study is to establish recommendations towards specific educational, preventative, rescue, or treatment strategies to reduce the number of fatal and non-fatal drowning incidents in Denmark (e.g., campaigns targeting high-risk groups, or fencing, allocating rescue equipment, or establishing lifeguard stations in high-risk areas).

Objectives

The primary objective is to estimate 30-day mortality of drowning incidents in Denmark treated by the Emergency Medical Services from 2016. The secondary objective is to explore risk factors associated with 30-day mortality.

Study design

A nationwide registry-based study linking data from the Danish Prehospital Drowning Data with data from the inhospital electronic medical records. from 2016 and follow-up on mortality 30 days after the drowning incident. Neurological outcomes will be assessed by trained observers through the inhospital electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Drowning
* Being registered in the Danish Prehospital Drowning Data with a valid civil registration number to allow for linkage with the inhospital electronic medical records

Exclusion Criteria:

* Obvious signs of irreversible death (decapitation, decomposition, post-mortem lividity, post-mortem rigidity).
* Declared dead on scene.
* A valid Do-Not-Attempt-Resuscitation order or other code status orders limiting life-sustaining therapies.
* An invalid civil registration number.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fatal and non-fatal drowning persons from 2016 identified in the Danish Prehospital Drowning Data.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days after the drowning incident
  The patient died before 30 days after the drowning incident
Neurological outcome | 30 days after the drowning incident
  Using the modified Ranking Scale (mRS) score

SECONDARY OUTCOMES:
Hospital length of stay | Immediately after hospital discharge
  Continuous
Intensive care unit admission | Immediately after hospital discharge
  Binary
Intensive care unit length of stay | Immediately after hospital discharge
  Continuous
Need for mechanical ventilation | Immediately after hospital discharge
  Binary
Duration of mechanical ventilation | Immediately after hospital discharge
  Continuous
Survival to hospital discharge | Immediately after hospital discharge
  Binary

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, Ass. Prof., Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center Region Zealand, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
Data are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Breindahl N, Wolthers SA, Jensen TW, Holgersen MG, Blomberg SNF, Steinmetz J, Christensen HC; Danish Cardiac Arrest Group. Danish Drowning Formula for identification of out-of-hospital cardiac arrest from drowning. Am J Emerg Med. 2023 Nov;73:55-62. doi: 10.1016/j.ajem.2023.08.024. Epub 2023 Aug 15. PMID 37619443